CLINICAL TRIAL: NCT03140332
Title: Contribution of the Perfusion Scanner in the Prediction of the Tumor Control of Patients With Hepatocellular Carcinoma Treated With Sorafenib.
Acronym: HCC-CTPerf
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PI2016_843_0025
Record Dates: First submitted 2017-04-27; First posted 2017-05-04 (Actual); Last update posted 2020-07-20 (Actual); Status verified 2020-07

CONDITIONS: Hepatocellular Carcinoma; Perfusion Scanner
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Therapeutics; Sorafenib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient with CHC (Other)
  Interventions: Other: Scannographic evaluation of the tumor response performed with mRECIST criteria after 3 months of treatment with sorafenib

INTERVENTIONS:
Other: Scannographic evaluation of the tumor response performed with mRECIST criteria after 3 months of treatment with sorafenib — To evaluate the association between tumor perfusion criteria (blood flow, blood volume, mean transit time, capillary permeability) at the initial perfusion scan and tumor control according to the mRECIST criteria after 3 months of treatment with sorafenib.

SUMMARY:
Hepatocellular carcinoma (HCC) is a hypervascular tumor. The reference treatment of advanced forms of stage C according to the Barcelona classification (BCLC C) is sorafenib, a multi-target tyrosine kinase inhibitor with predominant anti-angiogenic action. In order not to underestimate the efficacy of sorafenib, scannographic evaluation of the tumor response should be performed with mRECIST criteria that are significantly better correlated with survival. These criteria take into account the tumor size and also the modification of the tumor contrast enhancement after anti-angiogenic treatment. It seems appropriate to evaluate tumor control rather than tumor response since sorafenib is more stable than tumor response.

This evaluation will be made according to the mRECIST criteria after 3 months of treatment since the progression-free survival is of the order of 3 to 4 months. The determination of early predictive criteria for the response to sorafenib would optimize the management of advanced HCCs. Indeed, sorafenib only improves overall survival by 3 months in selected patients, and with undesirable effects and a significant cost. Predictive biological criteria have already been studied, such as alpha foeto-protein (AFP), whose early decrease with sorafenib is associated with better overall survival. The same applies to the early reduction at 4-6 weeks of tumor arterial contrast according to mRECIST criteria. The perfusion scanner appears to be an accessible and reproducible choice imaging technique for assessing tumor vasculature. In metastatic kidney cancers, it was demonstrated that some criteria for tumor perfusion prior to treatment with sorafenib were predictive of better control of the disease and even a better tumor response according to the RECIST 1.1 criteria. The determination of pre-therapeutic tumor perfusion criteria in order to predict tumor control or even overall survival has never been studied in advanced CHCs. On the other hand, an early variation in the criteria for tumor perfusion under treatment would tend to be correlated with the tumor response and even with overall progression-free survival.

Therefore, the study of tumor vascularization by the perfusion scanner could make it possible to demonstrate early predictive criteria for tumor control under sorafenib in order to optimize the management of patients with advanced HCC.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged over 18 years
* Affiliation to a social security scheme
* CHC developed irrespective of the level of fibrosis of the non-tumorous liver, and whatever the etiology
* Advanced hepatocellular carcinoma confirmed histologically or having the typical characteristics in imaging after validation in CPR (abdomino-pelvic CT scan with triphasic injection or hepatic MRI with gadolinium injection): hypervascularized nodule at the early arterial time (wash in) with washing ("Wash out") in relation to the non-tumoral parenchyma
* Hepatocellular carcinoma:

  * With a naive measurable target lesion of any treatment
  * Who can not benefit from curative treatment (non-operable, non-transplantable, non-radio-frequenable) and who have never benefited from systemic chemotherapy treatment
  * Or with appearance after chemo-embolization of target lesions according to the mRECIST criteria in the contralateral liver
* in the case of right or left arteriovenous fistula, the target lesion will be chosen in the contralateral liver
* Indication of treatment by sorafenib after validation in a multidisciplinary consultation meeting:

  * Stadium BCLC C
  * Cirrhosis classified Child-Pugh A or B7
  * Performance status less than or equal to 2
  * Preserved haematological function (platelet count ≥ 60000 / mm3, hemoglobin ≥ 8.5 g / dL)
  * Hepatic function (albumin ≥ 28 g / L, total bilirubin ≤ 50 μmol / L, ALAT and ASAT ≤ 5 N, INR ≤ 2.3 or TP> 40%)
  * Renal function conserved (creatinine ≤ 1.5 times the upper limit of normal)

Exclusion Criteria:

* Other evolutionary cancer requiring treatment
* History of treatment with sorafenib or anti-angiogenic therapy
* History of treatment by chemoembolization without appearance of target lesion in the contralateral liver
* Diffuse CHC with no measurable lesion
* Patient with TIPS, portal cavernoma, extensive portal thrombosis, or arterio-portal fistula in the same area of assessment of the CHC nodule
* Allergic reaction or hypersensitivity to a contrast agent
* Pregnancy
* Patient under tutorship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2017-02-27 (Actual); Primary Completion 2020-02-27 (Actual); Study Completion 2020-02-27 (Actual)

PRIMARY OUTCOMES:
Scannographic evaluation of tumor response with mRECIST criteria | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens Picardie, Amiens, Picardie, France